CLINICAL TRIAL: NCT03491267
Title: Pilot Exploratory Study to Determine Effect of Gentle Wounding to Stimulate Hair Follicle Neogenesis
Brief Title: Study to Determine Effect of Gentle Wounding to Stimulate Hair Follicle Neogenesis
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: National Institute Of Arthritis & Musculoskeletal & Skin Diseases (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: IRB00105061
Record Dates: First submitted 2018-03-23; First posted 2018-04-09 (Actual); Last update posted 2025-07-03 (Actual); Status verified 2025-07

CONDITIONS: Central Centrifugal Cicatricial Alopecia (CCCA)
Keywords: alopecia
MeSH Terms: conditions — Alopecia | interventions — Tretinoin; Lasers

STUDY DESIGN:
Intervention Model Description: Areas on a single scalp will be treated or untreated and monitored
Who Masked: Outcomes Assessor
Masking Description: assesors will be blinded
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Subjects with alopecia-- area treated (Experimental): One area will be treated
  Interventions: Drug: Retinoic acid; Device: Laser
- Subjects with alopecia-- area un-treated (Experimental): One area will be un-treated
  Interventions: Drug: Sham treatment; Device: Sham treatment

INTERVENTIONS:
Drug: Retinoic acid — The study team will treat skin with topical retinoic acid
  Arms: Subjects with alopecia-- area treated
Device: Laser — The study team treat skin with a surface laser.
  Arms: Subjects with alopecia-- area treated
Drug: Sham treatment — No drug will be given
  Arms: Subjects with alopecia-- area un-treated
Device: Sham treatment — No laser treatment will be given
  Arms: Subjects with alopecia-- area un-treated

SUMMARY:
The investigators have extensive evidence in mouse that wounding leads to the generation of new hair follicles in the skin. This can be an important new therapy for patients with scarring, but especially those with alopecia.

The question is whether gentle wounding in human subjects can cause the generation of a new hair follicle.

The plan is to first carefully map a small area of the scalp without hair follicles. Investigators will then try various modalities of gentle wounding (including fractionated Carbon Dioxide (CO2) laser, mild curetting) of the surface epithelium in the presence and absence of FDA approved topical medications (including retinoids). Investigators will then prospectively monitor the area for hair growth both by noninvasive visual monitoring (including photographs and dermoscopy) and biopsies.

The outcomes of this study hopefully will allow new therapies for especially scarring alopecia conditions where hair follicles are completely lost and there are no current therapies.

DETAILED DESCRIPTION:
Central centrifugal cicatricial alopecia (CCCA) is a scarring, inflammatory alopecia seen more commonly in women of African descent. The distinct pathophysiology of CCCA is poorly understood, but it is known to involve inflammation directed at the upper part of the hair follicle where the stem cells and sebaceous gland are located. If the stem cells and sebaceous gland are destroyed, there is no possibility for regeneration of the hair follicle, and permanent hair loss results. This form of scarring alopecia occurs mainly on the vertex of the scalp, and spreads peripherally, and can lead to baldness. In our dermatology clinics, our investigators see 5-10 patients per week for evaluation and treatment of CCCA.

Currently, treatment is focused on decreasing inflammation and halting the progression of disease. This typically consists of topical and intralesional corticosteroid therapy and anti-inflammatory antibiotics. Hair transplantation is the only treatment option for patients with end-stage CCCA, and has been performed in a small number of patients but the results have been disappointing with low graft survival rates and slow regrowth of the transplanted hair. In addition, hair transplantation of the curved hair follicles found in patients of African descent is difficult and requires specific expertise.

A study by Ito et al showed de novo hair follicle formation after wounding in genetically normal adult mice. The regenerated hair follicles were fully functional, in that they established a stem cell population, expressed known molecular markers of follicle differentiation, and produced a hair shaft that progressed normally through all stages of the hair follicle cycle. It is hypothesized that the regenerated hair follicles likely arise when epithelial cells in the wound assume a hair follicle stem cell phenotype, possibly under the influence of Wnt signaling.

The CO2 laser has been used extensively in dermatological surgery over the past 30 years and is now recognized as the gold standard for soft tissue vaporization. CO2 laser beam heats and vaporizes the skin tissue, instantly removing the superficial layers of the skin. Each fractional micro-spot creates a thermal zone. Intact cells around the treated area help during the healing process which in turn, induces cell regeneration. This likely occurs through dsRNA released during wounding. The investigators have recently found that retinoids, such as the tretinoin (retin-A) used in acne, can synergize with dsRNA and promote extra Wnt signaling.

The investigators therefore hypothesize that wounding of the area of scarring alopecia in CCCA, using a fractionated CO2 laser in combination with retinoid acid, will induce hair follicle regeneration.

ELIGIBILITY:
Inclusion criteria

Subjects who meet the following inclusion criteria will be included in the study:

* Male or female older than 18 at the screening visit;
* The subject is healthy, as determined by the investigator based on a medical evaluation including medical history;
* The subject has clinical diagnosis of CCCA;
* The subject's CCCA is of grades 2, 3 or 4, as assessed at the time of the screening visit.
* The subject is willing and able to comply with the requirements of the protocol. In particular, subject must adhere to the visits schedule, concomitant therapy and hair processing prohibitions, subject instructions, and biopsy procedures;
* The subject is willing to comply with the month long washout period if deemed necessary;
* The subject has understood and signed an Informed Consent Form approved by the Institutional Review Board (IRB) prior to any investigational procedure Exclusion criteria

Any subject who is meeting one or more of the following exclusion criteria at the screening visit and/or at the baseline visit will not be included in this study:

* The subject has an underlying known disease, a surgical or medical condition that in the opinion of the investigator might put the subject at risk
* The subject presents with any disease known or described to potentially interfere with a normal wound healing process
* The subject is pregnant or breastfeeding at the time of enrollment or is planning to become pregnant at any point during the study period (by self report)
* The subject has a past history of coagulation trouble
* The subject has a past history of abnormal healing (hypertrophic scars/keloids within the past 10 years)
* The subject has an underlying dermatological disease that in the opinion of the investigator could interfere with the study evaluations
* The subject has scars, sunburn, either damaged or broken (cuts or abrasions) skin or other blemishes, or tattoos on the scalp in the treatment area
* The subject is unwilling or unable to refrain from specific types of chemical hair styling and processing, including perms, straighteners, relaxers, dyes, weaves
* The subject has a known allergy or sensitivity to any local anesthetic drug (e.g. lidocaine) or a local antiseptic planned to be used for the laser and/or biopsy procedures
* The subject is in an exclusion period from a previous study or is participating in another clinical trial
* The subject is an adult under guardianship or is hospitalized in a public or private institution, or is deprived of freedom
* The subject is unable to communicate or cooperate with the Investigator due to language problems, poor mental development, or impaired cerebral function

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2024-11-01 (Actual); Study Completion 2024-11-01 (Actual)

PRIMARY OUTCOMES:
Hair follicle neogenesis as counted by in vivo scanning confocal microscopy | within 1 year of treatment
  appearance of new follicles, as defined by number of new follicles

CONTACTS AND LOCATIONS:
Overall Officials: Luis Garza, MD/PhD, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins School of Medicine, Dermatology Department, Baltimore, Maryland, United States